CLINICAL TRIAL: NCT04057183
Title: Noninvasive Evaluation for Carotid Artery Stenosis: The Carotid Stenotic Scan
Acronym: CSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phillip J Bendick (Industry)
Responsible Party: Sponsor-Investigator, Phillip J Bendick, Study Coordinator, CVR Medical
Organization: CVR Medical (Industry)
Other Study IDs: CVRMed
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Carotid Stenosis
Keywords: Carotid; Stenosis; Noninvasive
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Carotid Stenotic Scan — Noninvasive determination of presence or absence of carotid artery stenosis
  Other Names: CSS

SUMMARY:
The purpose of this study is to determine the accuracy of a new non-invasive device, the Carotid Stenotic Scan (CSS), to check for stenosis of the internal carotid artery (ICA) as compared to a carotid duplex ultrasound study.

DETAILED DESCRIPTION:
Currently, carotid duplex ultrasound is the primary diagnostic tool for the evaluation for ICA stenosis and must be performed by a trained and certified vascular technologist using advanced duplex imaging equipment and with subsequent interpretation by a trained physician. this test is not considered suitable for screening for disease. It would be of value to develop an accurate, reliable, low-cost, and easily accessible tool to screen for extra-cranial ICA disease in an office based setting. However, such a tool would require novel technology that allows for quick, accurate, reproducible, and safe evaluation.

This study will evaluate a new technology called the Carotid Stenotic Scan (CSS) developed by CVR Medical. The CSS instrument uses sensitive transducers to detect low frequency pressure fluctuations associated with flow disturbances downstream from areas of arterial narrowing.

Subjects will undergo a clinically ordered clinical carotid duplex ultrasound as part of standard of care. Subjects will have a noninvasive CSS assessment either before or after the carotid duplex ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 65 years scheduled for a diagnostic carotid artery duplex ultrasound study AND with one or more of the following:
* Hypertension
* Hyperlipidemia
* Diabetes
* Tobacco usage - Current or past
* Known CAD/PAD
* Family history of early onset of atherosclerotic disease

Exclusion Criteria:

* Unable / unwilling to provide Informed Consent
* Prior carotid endarterectomy or carotid artery stent
* Aortic stenosis
* Congestive heart failure
* BMI > 35

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Inclusion criteria identify an "at-risk" population with unknown carotid artery status. The literature indicates that patients who meet the criteria have a prevalence of significant carotid artery stenosis (>50%) of 7-10%. Current estimates are that 3 million adults in the United States have this degree of carotid artery disease with an annual stroke risk of 5-10%.
  Exclusion criteria are in place to identify patients in whom the status of the carotid arteries is already likely known (prior CEA or stent), have significant heart disease which will impact flow hemodynamics and create false negative or positive studies (CHF, aortic stenosis), or have excessive subcutaneous neck tissue that will attenuate and mask the CSS signal (elevated BMI).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of CSS result to carotid artery duplex ultrasound examination | CSS and duplex ultrasound done within one week of each other
  Percent agreement and negative predictive value of CSS compared to duplex ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Michigan Vascular Center, Flint, Michigan
  - Wake Forest Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared; only group data will be used.